CLINICAL TRIAL: NCT01877954
Title: Comparative Effectiveness of Extrafine Hydrofluoroalkane Beclometasone Versus Fluticasone in Paediatric Patients - a Retrospective, Real-life Observational Study in a uk Primary Care Asthma Population
Brief Title: Qvar vs FP in Pediatrics
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R02511
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: hydrofluoroalkane beclomethasone; fluticasone; paediatrics; real-life; observational; primary care
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IPDI Qvar: ICS initiation as Extra-fine hydrofluoroalkane beclometasone dipropionate
  Interventions: Drug: Extra-fine hydrofluoroalkane beclometasone dipropionate
- IPDI FP: ICS initiation as fluticasone propionate
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Extra-fine hydrofluoroalkane beclometasone dipropionate
  Other Names: Qvar®
  Groups: IPDI Qvar
Drug: Fluticasone propionate
  Groups: IPDI FP

SUMMARY:
The primary aim of this study was to compare the absolute and relative effectiveness of asthma management in paediatric patients in the UK on inhaled corticosteroid (ICS) maintenance therapy as extra-fine HFA-BDP (Qvar®) pressurised metered dose inhaler (pMDI) compared with fluticasone propionate (FP) pMDI.

DETAILED DESCRIPTION:
Comparison of asthma control with extrafine-particle hydrofluoroalkane-beclometasone (EF HFA-BDP) vs fluticasone propionate (FP) in paediatric patients (5-11year olds). Patients identified from the General Practice Research Database (GPRD) and the Optimum Patient Care Research Database (OPCRD). Two analyses were conducted:

1. Comparison of outcomes achieved by EF HFA-BDP and FP in 5-6year old patients with those achieved in 7-11yr old patients.
2. Comparison of outcomes achieved by EF HFA-BDP used with or without a spacer to those achieved by standard particle fluticasone propionate (FP) used with a spacer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged: 5-11 years
2. Evidence of asthma (diagnostic code and/or current asthma therapy);
3. Have at least one year of up-to-standard (UTS) baseline data (during which the step-up to FP/SAL occurred) and at least one year of UTS outcome data (following the IPD).

Exclusion Criteria:

1. Had any chronic respiratory disease, except asthma, at any time; and/or
2. Patients on maintenance oral steroids during baseline year

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Asthma patients who initiate ICS therapy as one of:
  HFA-BDP pMDI FP pMDI
Sampling Method: Non-Probability Sample
Enrollment: 2654 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Proxy risk domain asthma control | One year outcome period
  Defined as the absence of the following during the one-year outcome period:
  1. Asthma-related:
     * Hospital attendance or admission, OR
     * A&E attendance, OR
     * Out of hours attendance, OR
     * Out-patient department attendance
  2. GP consultations for lower respiratory tract infection
  3. Prescriptions for acute courses of oral steroids .
Asthma exacerbation rate ratio | One year outcome period
  Where exacerbations are defined as an occurrence of:
  Defined as an occurrence of:
  1. Asthma related:
     * Hospital admission, OR
     * A&E attendance, OR
  2. Use of acute oral steroids.

SECONDARY OUTCOMES:
Overall asthma control | One year outcome period
  Risk domain asthma control as defined above, plus
  (a)Average prescribed daily dose of albuterol or terbutaline of ≤200mg
Hospitalisation rates | One year outcome period
  Asthma-related hospitalisations
  1. Definite: Hospitalisations coded with an asthma read code
  2. Definite and probable: Hospitalisations with an asthma read code and uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of an asthma read code
  Respiratory hospitalisations
  1. Definite: Hospitalisations coded with a lower respiratory code
  2. Definite and probable: Hospitalisations with a lower respiratory read code and uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of a lower respiratory read code
Treatment success | One year outcome period
  Asthma control and no change in therapy
Adherence to ICS therapy | One year outcome period
  Categorised as: <50%, 50-<70%, 70-<100%, ≥100%.
Use of short-acting beta2-agonist ("reliever") therapy | One year outcome period

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Principal Investigator — Research in real life

REFERENCES:
- [Background] Leach CL, Davidson PJ, Hasselquist BE, Boudreau RJ. Influence of particle size and patient dosing technique on lung deposition of HFA-beclomethasone from a metered dose inhaler. J Aerosol Med. 2005 Winter;18(4):379-85. doi: 10.1089/jam.2005.18.379. PMID 16379614
- [Background] Leach CL, Davidson PJ, Boudreau RJ. Improved airway targeting with the CFC-free HFA-beclomethasone metered-dose inhaler compared with CFC-beclomethasone. Eur Respir J. 1998 Dec;12(6):1346-53. doi: 10.1183/09031936.98.12061346. PMID 9877489
- [Background] Giraud V, Roche N. Misuse of corticosteroid metered-dose inhaler is associated with decreased asthma stability. Eur Respir J. 2002 Feb;19(2):246-51. doi: 10.1183/09031936.02.00218402. PMID 11866004
- [Background] Newman SP, Weisz AW, Talaee N, Clarke SW. Improvement of drug delivery with a breath actuated pressurised aerosol for patients with poor inhaler technique. Thorax. 1991 Oct;46(10):712-6. doi: 10.1136/thx.46.10.712. PMID 1750017
- [Background] Newman SP, Millar AB, Lennard-Jones TR, Moren F, Clarke SW. Improvement of pressurised aerosol deposition with Nebuhaler spacer device. Thorax. 1984 Dec;39(12):935-41. doi: 10.1136/thx.39.12.935. PMID 6440305
- [Background] Chrystyn H, Price D. Not all asthma inhalers are the same: factors to consider when prescribing an inhaler. Prim Care Respir J. 2009 Dec;18(4):243-9. doi: 10.4104/pcrj.2009.00029. PMID 19513494
- [Background] Price D, Thomas M. Breaking new ground: challenging existing asthma guidelines. BMC Pulm Med. 2006 Nov 30;6 Suppl 1(Suppl 1):S6. doi: 10.1186/1471-2466-6-S1-S6. PMID 17140424
- [Result] Price D, Martin RJ, Barnes N, Dorinsky P, Israel E, Roche N, Chisholm A, Hillyer EV, Kemp L, Lee AJ, von Ziegenweidt J, Colice G. Prescribing practices and asthma control with hydrofluoroalkane-beclomethasone and fluticasone: a real-world observational study. J Allergy Clin Immunol. 2010 Sep;126(3):511-8.e1-10. doi: 10.1016/j.jaci.2010.06.040. Epub 2010 Aug 9. PMID 20692026